CLINICAL TRIAL: NCT01437514
Title: the Effect of the Preoperative Short-course Radiotherapy for the cT3/cN+ Mid-lower Rectal Cancer: a Prospective Randomized Study
Brief Title: Effective Study of Preoperative Short-course Radiotherapy for the Advanced Resectable Rectal Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ziqiang Wang,MD, associated professor of the West China Hospital, Sichuan University, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pSRT-201106
Record Dates: First submitted 2011-09-14; First posted 2011-09-21 (Estimated); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Rectal Neoplasms
Keywords: rectal cancer; Endosonography; preoperative short-course radiotherapy; preoperative adjuvant therapy; neoadjuvant therapy; short-term high-dose preoperative radiotherapy; total mesorectal excision; circumferential resection margin; local recurrence; overall survival; metastasis; complication
MeSH Terms: conditions — Rectal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- lower risk group with pSRT (Experimental): the patients that was divided into the lower risk group that the mesorectum involvement less than 5mm, and no lymph node larger than 8mm according to the preoperative CT, MRI and Endosonography,and these patients accept the preoperative short-course radiotherapy before the surgery
  Interventions: Radiation: preoperative short-course radiotherapy
- lower risk group with operation only (No Intervention): the patients that was divided into the lower risk group that the mesorectum involvement less than 5mm, and no lymph node larger than 8mm,according to the preoperative CT, MRI and Endosonography,and these patients have a operation directly without preoperative radiotherapy.
- higher risk group with pSRT (Experimental): the patients that was divided into the higher risk group that the mesorectum involvement more than 5mm, or with lymph node larger than 8mm according to the preoperative CT, MRI and Endosonography,and these patients have a operation directly without preoperative radiotherapy.these patients have the preoperative short-course radiotherapy before the surgery.
  Interventions: Radiation: preoperative short-course radiotherapy
- higher risk group with operation directly (No Intervention): the patients that was divided into the higher risk group that the mesorectum involvement more than 5mm, or with lymph node larger than 8mm according to the preoperative CT, MRI and Endosonography,and these patients have a operation directly without preoperative radiotherapy.

INTERVENTIONS:
Radiation: preoperative short-course radiotherapy — preoperative RT received a total dose of 25 Gy in five fractions during five consecutive days. The clinical target volume included the primary tumor and the mesentery with vascular supply containing the perirectal, presacral, and internal iliac nodes(up to the S1/S2 junction).The recommended upper border was at the level of the promontory. Radiation treatment was delivered with a three-portal technique.
  Other Names: short term regimen of high-dose preoperative radiotherapy (5×5 Gy); preoperative short term radiotherapy
  Arms: higher risk group with pSRT; lower risk group with pSRT

SUMMARY:
The local recurrence of rectal cancer is one of the main problem that fail the treatment. The preoperative neoadjuvant (chemo)radiotherapy has been confirmed to reduce the local recurrence rate,especially in the advanced rectal cancer. However the local recurrence rate is low about 10-20% totally,and the integrity of the mesorectum after the operation and circumferential resection margin(CRM) are the most critical factor for the local recurrence.So that, the advanced rectal cancer patients with negative CRM and had a complete mesorectum excision,may not benefit from the neoadjuvant radiation.This trial was mainly focus on the resectable advanced rectal cancer patients whose preoperative stage was cT3/N+. These patients will be divided into the lower risk group and higher risk group according the preoperative CT,Endoscopic ultrasound, and MRI,and carrying out randomized trial in the two groups respectively.The purpose of this trial is to confirm whether the preoperative radiotherapy is necessary for all the advanced rectal cancer patients,identify the reason of the local recurrence,and finally help the making of the treatment decision for the advanced resectable rectal cancer.

DETAILED DESCRIPTION:
The colorectal cancer is the secondary most common cancer among the population. Every year,it's estimated that there was over 1,200,000 new cases,and in China the data is about 440,000. The local recurrence (LR) and the lung or liver metastasis are the most critical problems that confusing the doctor,which the local recurrence rate is about 3%-50%,with a median rate of 18.8%。 Now, multidisciplinary treatment become a choice treatment for the rectal cancer, and the preoperative neoadjuvant (chemo)radiotherapy is a critical part of the treatment, as various trials have confirmed that the preoperative chemoradiotherapy can reduce the postoperative local recurrence rate. Although the preoperative radiotherapy can decrease the local recurrence, most of the studies show that it can't increase the overall survival. Also the large MRC study shows, the quality of operation is also critical for the local recurrence. and the main reasons of the local recurrence was thought to be the positive circumferential resection margin(CRM) and the remnant of the mesorectum. On the other hand, with the improvement of the TME surgery, the local recurrence of the advanced rectal cancer is lower than 20%, and the preoperative radiation may benefit half of these patients,and reduce the local recurrence rate to 7-10%.over 80% patients may be over treated and simultaneously suffer from the adverse effect of the radiation.The aim of this study was to explore that if the lower risk portion of the advanced rectal cancer patients is not necessary to have preoperative radiation,and the radiation will benefit the higher risk group.

In the trial,the operator will divide the resectable advanced rectal cancer patients (cT3/N+) into two subgroups according to the preoperative CT, MRI and EUS.firstly, the criteria of the lower risk group are: the tumor invade into the mesorectum<=5mm in lateral and posterior of the mesorectum, in the anterior wall the tumor had not invaded into the mesorectal fat tissue, there is no enlarged lymph node that larger than 8mm; and the higher risk group are: the tumor invade into the mesorectum >5mm in the lateral or posterior part, or invade into the mesorectum only in the anterior as the anterior mesorectum is relatively thin, or with lymph node larger than 8mm. then these patients were randomized to radiation with surgery or surgery only respectively. In the lower risk group we presume that the local recurrence rate is relatively low and the radiation can not improve LR, and in the higher risk group the radiation is significantly beneficial.

Of the preoperative radiation,there are two regimen,the long-term chemoradiotherapy and the short-course radiotherapy. mostly, the long-term regimen is more popular,with a total dose of 50.4 Gy in 25-28 fraction,compare to the short-term one with a dose of 25 Gy in 5 fraction, as the long-term regimen has a better effect of reduce the tumor invasion. For the resectable patients with negative CRM before the surgery,there is no conclusion which is better. so that the short-term radiation was choose as the regimen of this study.

Local recurrence after 3 years follow up has been chosen as primary endpoint. Proving a two-sided hypothesis of differences between the arms in higher risk group, the calculation of the sample size was based on expected local recurrence rates of 6% in the radiation group compared with 16% in the surgery group, resulting in altogether 210 patients (Log-Rank-test, with error of the 1st kind: α = 5% two-sided, power = 80%). As the lower risk group may have a very low LR rate, the totally 200 lower risk patients are planning to recruiting to randomization, which was similar to the higher risk group.

Patient baseline characteristics and disease factors were summarized using descriptive statistics. The categorical parameters were compared using two-sided Pearson's χ2 test or Fisher's exact test, as appropriate. All summary statistics on time-to-event variables were calculated according to the Kaplan-Meier method and were compared by means of the log-rank test. SPSS software(version 22.0; IBM, Chicago, IL) was used for statistical analyses. A P value<0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. histologically verified adenocarcinoma of the rectum;
2. the lower border of the tumor within 10cm of the anal verge;
3. age between 18 to 80 years;
4. preoperative endosonography,MRI and the abdominopelvic CT diagnosis as advanced rectal cancer (cT3/N+)(the detail of these two subgroup was illustrated in the detailed description of this trial);
5. ECOS ≤ 2
6. there was no evidence of metastasis with chest and abdominopelvic CT.

Exclusion Criteria:

1. with other colorectal cancer, or other cancer,simultaneously;
2. Locally recurrent rectal cancer;
3. had a history of malignant tumor within 5 years(except the skin cancer);
4. Pregnant or lactating women
5. there was contraindication for the preoperative adjuvant radiotherapy or the operation.
6. with antitumor drug or radiation before this trial.
7. discovery of metastasis in the operation
8. worrying about the local recurrence or the adverse effect of the radiation excessively;
9. with mental disorder.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2011-08; Primary Completion 2015-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
local recurrence | 3 years

SECONDARY OUTCOMES:
disease free survival | 3 years
  the time from operation to confirmed local recurrence, distant metastases, or death due to disease or treatment, whichever occurred first.
metastatic rate | 3 years
  ratio of the patients with metastasis after the operation
quality of life | 3 years
overall survival | 3 years
  the fraction of the person from the operation the death,no matter the reason of the death.
short-term complication of the surgery | first 30 day after operation

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Sichuan academy of medical science and sichuan provincial people's hospictal, Chengdu, Sichuan
  - the Third People'S Hospital of Chengdu, Chengdu, Sichuan
  - West China hospital, Sichuan University, Chengdu, Sichuan
  - The Third Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

REFERENCES:
- [Background] Korkolis DP, Plataniotis GD, Gondikakis E, Xinopoulos D, Koulaxouzidis GV, Katsilieris J, Vassilopoulos PP. Short-term preoperative radiotherapy is a safe approach for treatment of locally advanced rectal cancer. Int J Colorectal Dis. 2006 Jan;21(1):1-6. doi: 10.1007/s00384-005-0740-7. Epub 2005 Jun 10. PMID 15947936
- [Background] Gu J, Wang L. [Standardized examination and research advancement of circumferential resection margin in patients with middle-lower rectal cancer]. Zhonghua Wei Chang Wai Ke Za Zhi. 2011 Apr;14(4):229-33. Chinese. PMID 21538262
- [Background] Frasson M, Garcia-Granero E, Roda D, Flor-Lorente B, Rosello S, Esclapez P, Faus C, Navarro S, Campos S, Cervantes A. Preoperative chemoradiation may not always be needed for patients with T3 and T2N+ rectal cancer. Cancer. 2011 Jul 15;117(14):3118-25. doi: 10.1002/cncr.25866. Epub 2011 Jan 24. PMID 21264832
- [Background] Stephens RJ, Thompson LC, Quirke P, Steele R, Grieve R, Couture J, Griffiths GO, Sebag-Montefiore D. Impact of short-course preoperative radiotherapy for rectal cancer on patients' quality of life: data from the Medical Research Council CR07/National Cancer Institute of Canada Clinical Trials Group C016 randomized clinical trial. J Clin Oncol. 2010 Sep 20;28(27):4233-9. doi: 10.1200/JCO.2009.26.5264. Epub 2010 Jun 28. PMID 20585099
- [Background] Kav T, Bayraktar Y. How useful is rectal endosonography in the staging of rectal cancer? World J Gastroenterol. 2010 Feb 14;16(6):691-7. doi: 10.3748/wjg.v16.i6.691. PMID 20135716
- [Background] Pietrzak L, Bujko K, Nowacki MP, Kepka L, Oledzki J, Rutkowski A, Szmeja J, Kladny J, Dymecki D, Wieczorek A, Pawlak M, Lesniak T, Kowalska T, Richter P; Polish Colorectal Study Group. Quality of life, anorectal and sexual functions after preoperative radiotherapy for rectal cancer: report of a randomised trial. Radiother Oncol. 2007 Sep;84(3):217-25. doi: 10.1016/j.radonc.2007.07.007. Epub 2007 Aug 10. PMID 17692977
- [Background] Peeters KC, Marijnen CA, Nagtegaal ID, Kranenbarg EK, Putter H, Wiggers T, Rutten H, Pahlman L, Glimelius B, Leer JW, van de Velde CJ; Dutch Colorectal Cancer Group. The TME trial after a median follow-up of 6 years: increased local control but no survival benefit in irradiated patients with resectable rectal carcinoma. Ann Surg. 2007 Nov;246(5):693-701. doi: 10.1097/01.sla.0000257358.56863.ce. PMID 17968156
- [Background] van Gijn W, Marijnen CA, Nagtegaal ID, Kranenbarg EM, Putter H, Wiggers T, Rutten HJ, Pahlman L, Glimelius B, van de Velde CJ; Dutch Colorectal Cancer Group. Preoperative radiotherapy combined with total mesorectal excision for resectable rectal cancer: 12-year follow-up of the multicentre, randomised controlled TME trial. Lancet Oncol. 2011 Jun;12(6):575-82. doi: 10.1016/S1470-2045(11)70097-3. Epub 2011 May 17. PMID 21596621
- [Background] Kapiteijn E, Marijnen CA, Nagtegaal ID, Putter H, Steup WH, Wiggers T, Rutten HJ, Pahlman L, Glimelius B, van Krieken JH, Leer JW, van de Velde CJ; Dutch Colorectal Cancer Group. Preoperative radiotherapy combined with total mesorectal excision for resectable rectal cancer. N Engl J Med. 2001 Aug 30;345(9):638-46. doi: 10.1056/NEJMoa010580. PMID 11547717
- [Background] Sebag-Montefiore D, Stephens RJ, Steele R, Monson J, Grieve R, Khanna S, Quirke P, Couture J, de Metz C, Myint AS, Bessell E, Griffiths G, Thompson LC, Parmar M. Preoperative radiotherapy versus selective postoperative chemoradiotherapy in patients with rectal cancer (MRC CR07 and NCIC-CTG C016): a multicentre, randomised trial. Lancet. 2009 Mar 7;373(9666):811-20. doi: 10.1016/S0140-6736(09)60484-0. PMID 19269519
- [Background] Swedish Rectal Cancer Trial; Cedermark B, Dahlberg M, Glimelius B, Pahlman L, Rutqvist LE, Wilking N. Improved survival with preoperative radiotherapy in resectable rectal cancer. N Engl J Med. 1997 Apr 3;336(14):980-7. doi: 10.1056/NEJM199704033361402. PMID 9091798
- [Background] Folkesson J, Birgisson H, Pahlman L, Cedermark B, Glimelius B, Gunnarsson U. Swedish Rectal Cancer Trial: long lasting benefits from radiotherapy on survival and local recurrence rate. J Clin Oncol. 2005 Aug 20;23(24):5644-50. doi: 10.1200/JCO.2005.08.144. PMID 16110023
- [Background] Birgisson H, Pahlman L, Gunnarsson U, Glimelius B; Swedish Rectal Cancer Trial Group. Adverse effects of preoperative radiation therapy for rectal cancer: long-term follow-up of the Swedish Rectal Cancer Trial. J Clin Oncol. 2005 Dec 1;23(34):8697-705. doi: 10.1200/JCO.2005.02.9017. PMID 16314629
- [Derived] Deng X, Liu P, Jiang D, Wei M, Wang X, Yang X, Zhang Y, Wu B, Liu Y, Qiu M, Zhuang H, Zhou Z, Li Y, Xu F, Wang Z. Neoadjuvant Radiotherapy Versus Surgery Alone for Stage II/III Mid-low Rectal Cancer With or Without High-risk Factors: A Prospective Multicenter Stratified Randomized Trial. Ann Surg. 2020 Dec;272(6):1060-1069. doi: 10.1097/SLA.0000000000003649. PMID 31599809